CLINICAL TRIAL: NCT00910065
Title: A Prospective, Randomized, Verum Controlled, Open Label, Parallel Group Multi-center Phase III Clinical Trial to Demonstrate the Superiority of 500 or 250 mg Aspirin® i.v. (BAY 81-8781) Treatment Versus 300 mg Aspirin® N Tablets p.o. (BAY e4465A) in Patients With Acute Coronary Syndrome, Measured by Time Dependent Thromboxane Inhibition
Brief Title: BAY81-8781, I.V. Aspirin in the Indication of Acute Coronary Syndrome (ACS)
Acronym: ACUTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12946; 2007-005163-94 (EudraCT Number)
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; ACS; Aspirin
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: D,L-lysine acetylsalicylate (Aspirin, BAY81-8781) 500 mg IV
- Arm 2 (Experimental)
  Interventions: Drug: D,L-lysine acetylsalicylate (Aspirin, BAY81-8781) 250 mg IV
- Arm 3 (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYe4465) 300 mg Tablet

INTERVENTIONS:
Drug: D,L-lysine acetylsalicylate (Aspirin, BAY81-8781) 500 mg IV — Single IV dose of aspirin at a dose of 500 mg as bolus infusion injection in approximately 30 seconds through the vein on Day 1.
  Arms: Arm 1
Drug: D,L-lysine acetylsalicylate (Aspirin, BAY81-8781) 250 mg IV — Single IV dose of aspirin at a dose of 250 mg as bolus infusion injection in approximately 30 seconds through the vein on Day 1.
  Arms: Arm 2
Drug: Acetylsalicylic acid (Aspirin, BAYe4465) 300 mg Tablet — Single oral dose of aspirin tablet at a dose of 300 mg on Day 1.
  Arms: Arm 3

SUMMARY:
The objective of this study is to investigate whether intravenous administration (injected into a vein) of acetylsalicylic acid (Aspirin) in doses of 250 and 500 mg is superior to oral treatment of ACS with tablets containing 300 mg of Aspirin.

DETAILED DESCRIPTION:
In November 2009 it was the company's decision to cancel this study as an international trial. However, to support the local MA application of Aspirin i.v. for the indication "For the initial treatment in case of suspicion of acute coronary syndrome", Bayer decided to perform this trial in Germany as a domestic trial, with changed number of participants and study dates.

ELIGIBILITY:
Inclusion Criteria:

* Angina pectoris lasting for more than 20 minutes within the last 24 hours before study drug treatment (or equivalent acute symptoms such as increasing dyspnea, diaphoresis, nausea, abdominal/epigastric pain, syncope etc.)
* ECG change suggestive for ischemia:
* ST elevation or T-wave change or ST depression, new or presumed left bundle-branch block (LBBB)
* Elevated troponin T level > 0.01 ng/ml, levels according to local laboratory reference values
* Risk factors for ACS such as known coronary artery disease (CAD), diabetes mellitus, impaired renal function, peripheral artery or cerebrovascular disease, current smoking.

Exclusion Criteria:

* Treatment with acetylsalicylic acid (ASA) within 48 hours prior to study drug treatment
* Treatment with glycoprotein IIa/IIIb inhibitors within 48 hours prior to study drug treatment and before the 20 minutes blood samples for thromboxane, prostacycline and platelet aggregation measurement have been taken
* Thrombolytic therapy within 24 hours before study drug treatment
* Obligation for tracheal intubation and mechanical ventilation
* Contraindications to ASA treatment
* Known haemorrhagic diathesis
* Evidence of an active gastrointestinal or urogenital bleeding
* Stroke within 3 months prior to study drug treatment
* Major surgery including coronary artery bypass graft (CABG) within 6 weeks prior to study drug treatment
* Known severe hepatic or renal insufficiency
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Concentration of Thromboxane B2 (TXB2) at 5 Minutes Post-dose | 5 minutes post-dose

SECONDARY OUTCOMES:
Concentration of Thromboxane B2 (TXB2) at 20 Minutes Post-dose | 20 minutes post-dose
Platelet Aggregation Inhibition (PAI) at 5 Minutes and 20 Minutes After Single Dose of Study Drug Administration Measured as Response to Treatment | 5 and 20 minutes post-dose
Serum Concentration of Prostacyclin Metabolite at 5 and 20 Minutes Post-dose | 5 and 20 minutes post-dose
Incidence of the Composite Clinical Endpoint of Cardiovascular Death, Stroke and Myocardial Infarction up to Day 30 After Single Dose of Study Drug Administration | Post-randomization up to 30 days after single dose of study drug administration
Incidence of Post-randomization Deaths From all Causes, Cardiovascular Deaths, Myocardial Re/Infarctions and Ischemic Strokes Within 24 Hours, 7 Days And 30 Days After Single Dose of Study Drug Administration | Post-randomization up to 24 hours, 7 days and 30 days after single dose of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- China (7):
  - Guangzhou, Guangdong
  - Changsha, Hunan
  - Nanchang, Jiangxi
  - Shenyang, Liaoning
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
- Germany (15):
  - Bad Krozingen, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Coburg, Bavaria
  - Dachau, Bavaria
  - Melsungen, Hesse
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Soest, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Worms, Rhineland-Palatinate
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Moscow, Russia
- Spain (4):
  - Alicante, Alicante
  - San Juan, Alicante
  - Sabadell, Barcelona
  - Valencia, Valencia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/